CLINICAL TRIAL: NCT06599216
Title: Adebrelimab Combined With Dalpicicliband Standard Endocrine Therapy for HR + / HER 2-breast Cancer:A Single-center,Open-label,Single-arm Clinical Trial
Brief Title: Adebrelimab Combined With Dalpiciclib and Standard Endocrine Therapy for HR + / HER2- Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Jinsong Wang, Professor of Treatment, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-071
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; HR+/HER2- Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Adebrelimab+Dalpciclib+Standard Endocrine Therapy

INTERVENTIONS:
Drug: Adebrelimab+Dalpciclib+Standard Endocrine Therapy — Adebrelimab: 1200mg, intravenously, Q4w Dalpiciclib: 150mg once a day for 3 weeks, stop for 1 week, Q4w Standard Endocrine Therapy: Choice of endocrine therapy is according to guidelines and centre policy by investigator

SUMMARY:
This study intends to explore the efficacy and safety of PD-L1 inhibitor Adebrelimab combined with the CDK4/6 inhibitor Dalpcicilib and standard endocrine therapy given as neoadjuvant treatment in stages II-III hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer.

DETAILED DESCRIPTION:
This single-center, open-label, single-arm clinical trial aims to evaluate the efficacy and safety of the neoadjuvant treatment with the PD-L1 inhibitor Adebrelimab in combination with the CDK4/6 inhibitor Dalpicicilib in combination with standard endocrine therapy, for stages II-III hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women, aged ≥18 years;
2. Postmenopausal patients and all patients in the screening period must one of the following:

   * Previous bilateral oophorectomy, or aged ≥60 years;
   * Aged <60 years, natural Postmenopausal status (defined as spontaneous cessation for at least 12 consecutive months without other pathological or physiological causes), E2 and FSH at the postmenopausal level;
3. Histologically confirmed HR+/HER2- invasive breast cancer (specific definition: ER >10% tumor cell positive is defined as ER positive, PR >10% tumor cell positive is defined as PR positive, ER and/or PR positive is defined as HR positive; HER2 0-1+ or HER2 ++ but negative by FISH test, no amplification, defined as HER2 negative);
4. Histologically confirmed invasive breast cancer, stage II-III breast cancer diagnosed based on AJCC cancer staging system (8th edition) ;
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
6. According to the RECIST 1.1 standard, at least one measurable lesion exists;
7. The main organs have basically normal functions and meet the following conditions:

   * Bone marrow function: Hb≥90 g/L (no blood was transfused within 14 days); ANC≥1.5×109/L;PLT≥80×I09/L;
   * Liver and kidney function: TBlL≤1.5×ULN; ALT and AST≤3×ULN; serum Cr≤1.5 ULN and creatinine clearance>50 ml/min (Cockcroft-Gault formula);
8. Subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Previous use of CDK4/6 inhibitors or PD1/PD-L1 monoclonal antibody or concurrent treatment with any other antitumor therapy;
2. Severe organ dysfunction;
3. Inability to swallow,chronic diarrhea and intestinal obstruction,there are multiple factors that affect drug intake and absorption;
4. Patients with known HBV or HCV infection active phase or HBV DNA≥500, or chronic phase with abnormal liver function;
5. History of active autoimmune disease (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes)
6. History of immunodeficiency, including HIV testing positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation; History of interstitial lung disease (except radiation pneumonia without hormone therapy) and non-infectious pneumonia;
7. History of any heart disease, including:1)medicated or clinically significant arrhythmia; 2) myocardial infarction; 3) heart failure; 4) any other cardiac disease judged by the investigator for the trial;
8. Patients during pregnancy and lactation, women of childbearing age who refuse to take effective contraceptive measures during the study period;
9. According to the discretion of the investigator, there are significant risks to patient safety or concomitant diseases affecting the patient's completion of the study (including but not limited to severe hypertension, severe diabetes, active infection);
10. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia;
11. Any condition deemed inappropriate for the patient's participation in this study by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
tpCR rate | through study completion, an average of one and a half years
  Total pathologic complete response (tpCR) rate, defined as ypT0/is, ypN0 as assessed by investigator.

SECONDARY OUTCOMES:
OS | up to 3 years
  OS is defined as the time between enrollment and the patient's death due to any cause.
EFS | up to 3 years
  Event-Free Survival (EFS) is defined as the time from firest dose to disease progression, disease recurrence, or death, whichever comes first.
Ki67 | Baseline and At Surgery
  Evaluation by a pathologist by manual counting according to WHO 2017 recommendations
ORR | Baseline up to Cycle 5（each cycle is 28 days）
  Objective response rate(ORR) is defined as the proportion of patients with complete response(CR) and partial response(PR) assessed by the investigator in accordance with the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical Cancer Hospital, Harbin, Heilongjiang
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang P, Zhang Q, Tong Z, Sun T, Li W, Ouyang Q, Hu X, Cheng Y, Yan M, Pan Y, Teng Y, Yan X, Wang Y, Xie W, Zeng X, Wang X, Hu C, Geng C, Zhang H, Li W, Wu X, Zhong J, Xu J, Shi Y, Wei W, Bayaxi N, Zhu X, Xu B. Dalpiciclib plus letrozole or anastrozole versus placebo plus letrozole or anastrozole as first-line treatment in patients with hormone receptor-positive, HER2-negative advanced breast cancer (DAWNA-2): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2023 Jun;24(6):646-657. doi: 10.1016/S1470-2045(23)00172-9. Epub 2023 May 11. PMID 37182538
- [Background] Xu B, Zhang Q, Zhang P, Hu X, Li W, Tong Z, Sun T, Teng Y, Wu X, Ouyang Q, Yan X, Cheng J, Liu Q, Feng J, Wang X, Yin Y, Shi Y, Pan Y, Wang Y, Xie W, Yan M, Liu Y, Yan P, Wu F, Zhu X, Zou J; DAWNA-1 Study Consortium. Dalpiciclib or placebo plus fulvestrant in hormone receptor-positive and HER2-negative advanced breast cancer: a randomized, phase 3 trial. Nat Med. 2021 Nov;27(11):1904-1909. doi: 10.1038/s41591-021-01562-9. Epub 2021 Nov 4. PMID 34737452
- [Background] Wang J, Zhou C, Yao W, Wang Q, Min X, Chen G, Xu X, Li X, Xu F, Fang Y, Yang R, Yu G, Gong Y, Zhao J, Fan Y, Liu Q, Cao L, Yao Y, Liu Y, Li X, Wu J, He Z, Lu K, Jiang L, Hu C, Zhao W, Zhang B, Shi W, Zhang X, Cheng Y; CAPSTONE-1 Study Group. Adebrelimab or placebo plus carboplatin and etoposide as first-line treatment for extensive-stage small-cell lung cancer (CAPSTONE-1): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Jun;23(6):739-747. doi: 10.1016/S1470-2045(22)00224-8. Epub 2022 May 13. PMID 35576956
- [Background] Nanda R, Liu MC, Yau C, Shatsky R, Pusztai L, Wallace A, Chien AJ, Forero-Torres A, Ellis E, Han H, Clark A, Albain K, Boughey JC, Jaskowiak NT, Elias A, Isaacs C, Kemmer K, Helsten T, Majure M, Stringer-Reasor E, Parker C, Lee MC, Haddad T, Cohen RN, Asare S, Wilson A, Hirst GL, Singhrao R, Steeg K, Asare A, Matthews JB, Berry S, Sanil A, Schwab R, Symmans WF, van 't Veer L, Yee D, DeMichele A, Hylton NM, Melisko M, Perlmutter J, Rugo HS, Berry DA, Esserman LJ. Effect of Pembrolizumab Plus Neoadjuvant Chemotherapy on Pathologic Complete Response in Women With Early-Stage Breast Cancer: An Analysis of the Ongoing Phase 2 Adaptively Randomized I-SPY2 Trial. JAMA Oncol. 2020 May 1;6(5):676-684. doi: 10.1001/jamaoncol.2019.6650. PMID 32053137
- [Background] Tolaney SM, Barroso-Sousa R, Keenan T, Li T, Trippa L, Vaz-Luis I, Wulf G, Spring L, Sinclair NF, Andrews C, Pittenger J, Richardson ET 3rd, Dillon D, Lin NU, Overmoyer B, Partridge AH, Van Allen E, Mittendorf EA, Winer EP, Krop IE. Effect of Eribulin With or Without Pembrolizumab on Progression-Free Survival for Patients With Hormone Receptor-Positive, ERBB2-Negative Metastatic Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1598-1605. doi: 10.1001/jamaoncol.2020.3524. PMID 32880602
- [Background] Rugo HS, Delord JP, Im SA, Ott PA, Piha-Paul SA, Bedard PL, Sachdev J, Le Tourneau C, van Brummelen EMJ, Varga A, Salgado R, Loi S, Saraf S, Pietrangelo D, Karantza V, Tan AR. Safety and Antitumor Activity of Pembrolizumab in Patients with Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer. Clin Cancer Res. 2018 Jun 15;24(12):2804-2811. doi: 10.1158/1078-0432.CCR-17-3452. Epub 2018 Mar 20. PMID 29559561
- [Background] Dieci MV, Griguolo G, Miglietta F, Guarneri V. The immune system and hormone-receptor positive breast cancer: Is it really a dead end? Cancer Treat Rev. 2016 May;46:9-19. doi: 10.1016/j.ctrv.2016.03.011. Epub 2016 Mar 28. PMID 27055087
- [Background] Johnston SR, Kilburn LS, Ellis P, Dodwell D, Cameron D, Hayward L, Im YH, Braybrooke JP, Brunt AM, Cheung KL, Jyothirmayi R, Robinson A, Wardley AM, Wheatley D, Howell A, Coombes G, Sergenson N, Sin HJ, Folkerd E, Dowsett M, Bliss JM; SoFEA investigators. Fulvestrant plus anastrozole or placebo versus exemestane alone after progression on non-steroidal aromatase inhibitors in postmenopausal patients with hormone-receptor-positive locally advanced or metastatic breast cancer (SoFEA): a composite, multicentre, phase 3 randomised trial. Lancet Oncol. 2013 Sep;14(10):989-98. doi: 10.1016/S1470-2045(13)70322-X. Epub 2013 Jul 29. PMID 23902874
- [Background] Prat A, Saura C, Pascual T, Hernando C, Munoz M, Pare L, Gonzalez Farre B, Fernandez PL, Galvan P, Chic N, Gonzalez Farre X, Oliveira M, Gil-Gil M, Arumi M, Ferrer N, Montano A, Izarzugaza Y, Llombart-Cussac A, Bratos R, Gonzalez Santiago S, Martinez E, Hoyos S, Rojas B, Virizuela JA, Ortega V, Lopez R, Celiz P, Ciruelos E, Villagrasa P, Gavila J. Ribociclib plus letrozole versus chemotherapy for postmenopausal women with hormone receptor-positive, HER2-negative, luminal B breast cancer (CORALLEEN): an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2020 Jan;21(1):33-43. doi: 10.1016/S1470-2045(19)30786-7. Epub 2019 Dec 11. PMID 31838010
- [Background] Cottu P, D'Hondt V, Dureau S, Lerebours F, Desmoulins I, Heudel PE, Duhoux FP, Levy C, Mouret-Reynier MA, Dalenc F, Frenel JS, Jouannaud C, Venat-Bouvet L, Nguyen S, Ferrero JM, Canon JL, Grenier J, Callens C, Gentien D, Lemonnier J, Vincent-Salomon A, Delaloge S. Letrozole and palbociclib versus chemotherapy as neoadjuvant therapy of high-risk luminal breast cancer. Ann Oncol. 2018 Dec 1;29(12):2334-2340. doi: 10.1093/annonc/mdy448. PMID 30307466
- [Background] Hurvitz SA, Martin M, Press MF, Chan D, Fernandez-Abad M, Petru E, Rostorfer R, Guarneri V, Huang CS, Barriga S, Wijayawardana S, Brahmachary M, Ebert PJ, Hossain A, Liu J, Abel A, Aggarwal A, Jansen VM, Slamon DJ. Potent Cell-Cycle Inhibition and Upregulation of Immune Response with Abemaciclib and Anastrozole in neoMONARCH, Phase II Neoadjuvant Study in HR+/HER2- Breast Cancer. Clin Cancer Res. 2020 Feb 1;26(3):566-580. doi: 10.1158/1078-0432.CCR-19-1425. Epub 2019 Oct 15. PMID 31615937
- [Background] Ma CX, Gao F, Luo J, Northfelt DW, Goetz M, Forero A, Hoog J, Naughton M, Ademuyiwa F, Suresh R, Anderson KS, Margenthaler J, Aft R, Hobday T, Moynihan T, Gillanders W, Cyr A, Eberlein TJ, Hieken T, Krontiras H, Guo Z, Lee MV, Spies NC, Skidmore ZL, Griffith OL, Griffith M, Thomas S, Bumb C, Vij K, Bartlett CH, Koehler M, Al-Kateb H, Sanati S, Ellis MJ. NeoPalAna: Neoadjuvant Palbociclib, a Cyclin-Dependent Kinase 4/6 Inhibitor, and Anastrozole for Clinical Stage 2 or 3 Estrogen Receptor-Positive Breast Cancer. Clin Cancer Res. 2017 Aug 1;23(15):4055-4065. doi: 10.1158/1078-0432.CCR-16-3206. Epub 2017 Mar 7. PMID 28270497
- [Background] Johnston S, Puhalla S, Wheatley D, Ring A, Barry P, Holcombe C, Boileau JF, Provencher L, Robidoux A, Rimawi M, McIntosh SA, Shalaby I, Stein RC, Thirlwell M, Dolling D, Morden J, Snowdon C, Perry S, Cornman C, Batten LM, Jeffs LK, Dodson A, Martins V, Modi A, Osborne CK, Pogue-Geile KL, Cheang MCU, Wolmark N, Julian TB, Fisher K, MacKenzie M, Wilcox M, Huang Bartlett C, Koehler M, Dowsett M, Bliss JM, Jacobs SA. Randomized Phase II Study Evaluating Palbociclib in Addition to Letrozole as Neoadjuvant Therapy in Estrogen Receptor-Positive Early Breast Cancer: PALLET Trial. J Clin Oncol. 2019 Jan 20;37(3):178-189. doi: 10.1200/JCO.18.01624. Epub 2018 Dec 6. PMID 30523750
- [Background] Spring LM, Fell G, Arfe A, Sharma C, Greenup R, Reynolds KL, Smith BL, Alexander B, Moy B, Isakoff SJ, Parmigiani G, Trippa L, Bardia A. Pathologic Complete Response after Neoadjuvant Chemotherapy and Impact on Breast Cancer Recurrence and Survival: A Comprehensive Meta-analysis. Clin Cancer Res. 2020 Jun 15;26(12):2838-2848. doi: 10.1158/1078-0432.CCR-19-3492. Epub 2020 Feb 11. PMID 32046998
- [Background] Cejalvo JM, Pascual T, Fernandez-Martinez A, Braso-Maristany F, Gomis RR, Perou CM, Munoz M, Prat A. Clinical implications of the non-luminal intrinsic subtypes in hormone receptor-positive breast cancer. Cancer Treat Rev. 2018 Jun;67:63-70. doi: 10.1016/j.ctrv.2018.04.015. Epub 2018 May 7. PMID 29763779
- [Background] Goel S, Bergholz JS, Zhao JJ. Targeting CDK4 and CDK6 in cancer. Nat Rev Cancer. 2022 Jun;22(6):356-372. doi: 10.1038/s41568-022-00456-3. Epub 2022 Mar 18. PMID 35304604
- [Background] Geum D, Sun W, Paik SK, Lee CC, Kim K. Estrogen-induced cyclin D1 and D3 gene expressions during mouse uterine cell proliferation in vivo: differential induction mechanism of cyclin D1 and D3. Mol Reprod Dev. 1997 Apr;46(4):450-8. doi: 10.1002/(SICI)1098-2795(199704)46:43.0.CO;2-N. PMID 9094091
- [Background] Pernas S, Tolaney SM, Winer EP, Goel S. CDK4/6 inhibition in breast cancer: current practice and future directions. Ther Adv Med Oncol. 2018 Jul 17;10:1758835918786451. doi: 10.1177/1758835918786451. eCollection 2018. PMID 30038670
- [Background] Spring LM, Gupta A, Reynolds KL, Gadd MA, Ellisen LW, Isakoff SJ, Moy B, Bardia A. Neoadjuvant Endocrine Therapy for Estrogen Receptor-Positive Breast Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1477-1486. doi: 10.1001/jamaoncol.2016.1897. PMID 27367583